CLINICAL TRIAL: NCT05394506
Title: Identification of Genetic Modifying Factors in Striated Muscle Laminopathies
Brief Title: Modifying Factors in Striated Muscle Laminopathies
Acronym: LMNAModifier
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C20-45
Record Dates: First submitted 2022-03-30; First posted 2022-05-27 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Laminopathies; Emery Dreifuss Muscular Dystrophy 2; LMNA-Related Congenital Muscular Dystrophy; Dilated Cardiomyopathy-1A
Keywords: A-type lamins; LMNA; muscular dystrophy; modifier factor
MeSH Terms: conditions — Laminopathies; Autosomal Emery-Dreifuss Muscular Dystrophy; Muscular Dystrophy, Congenital, Lmna-Related; Cardiomyopathy, Dilated; Muscular Dystrophies

STUDY DESIGN:
Intervention Model Description: * To collect biological material (muscle and/or skin biopsies) and the phenotype of patients with mutations in the LMNA gene (within large families with variable clinical presentation or within cohorts of patients with recurrent mutations in the LMNA gene.
  * To grade the severity of the muscle phenotype of these patients (severe, moderate, mild).
  * Perform "omics" analysis on their biological material.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collection of biological material (Other): Patients carrying LMNA mutation with no contrindication for skin and/or muscle biopsy:
  * from large families with striking intrafamilial phenotypic variability (3 families identified).
  * patients carrying p.Arg453Trp or p.Glu358Lys LMNA gene mutations
  Interventions: Procedure: Skin Biopsy; Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Skin Biopsy — The skin biopsy is performed in the consultation outclinic room. A local anaesthetic (anaesthetic patch to be applied to the skin) is required for this procedure. The skin biopsy is usually performed on the front of the forearm (but can be performed on the arm, thigh or leg). After disinfection, a fragment of 3 to 4 mm in diameter is removed with a biopsy-punch (single-use device). If necessary, a suture can be placed. Otherwise, the wound is covered with Steristrip and a sterile dressing. The skin sample, intended for a fibroblast culture, will be placed in a flask to be kept at room temperature. It will be labelled with specific labels and sent to the local biological resource centre.
Procedure: Muscle biopsy — The muscle biopsy is performed in a sterile room. A local anaesthetic is required for this procedure. After selecting the muscle from which the sample will be taken (usually from the deltoid muscle at the shoulder stump), placing a sterile field and disinfecting, a small incision is made in the skin until the selected muscle is exposed. A bundle of muscle fibres of approximately 1 cm x 0.5 cm is removed. The skin is then sutured and covered with a sterile dressing. The procedure takes about 30 minutes (including patient set-up). The muscle sample will be divided into 2 fragments, one for myoblast culture, the other for frozen tissue. The 2 vials will be labelled with specific labels and then sent to the local biological resource centre

SUMMARY:
Mutations in the LMNA gene, which codes for lamins A and C, proteins of the nuclear lamina, are responsible for a wide spectrum of pathologies, including a group specifically affecting striated skeletal and cardiac muscles, with cardiac involvement being life-threatening. At the skeletal muscle level, a wide phenotypic spectrum has been described, ranging from severe forms of congenital muscular dystrophy to less severe forms of limb-girdle muscular dystrophy. The great clinical variability of striated muscle laminopathies, both inter- and intra-familial, can be observed in the age of onset, severity of signs and progression of muscle and heart involvement. To date, more than 400 LMNA mutations have been associated with striated muscle laminopathies (www.umd.be/LMNA/), highlighting strong clinical and genetic heterogeneity. A few recurrent mutations linked to a difference in severity have been identified. However, these genotype-phenotype relationships and the rare cases of digenism reported do not explain all the clinical variability of laminopathies. Therefore, there are probably other factors of severity than the causative mutation, called "modifier genes".

Identification of such modifier genes has been initiated by studying a large family with significant clinical variability in the age of onset of muscle signs. A segregation analysis within this family identified 2 potential modifier loci. High-throughput sequencing restricted to these 2 regions according to phenotypic subgroups did not led to meaningful results so far. In addition, an international retrospective study of the natural history of early muscle laminopathies has allowed the investigators to highlight a strong inter-family clinical variability in patients carrying recurrent mutations. The investigators thus have strong preliminary data that could allow them to identify modifying genetic factors in a cohort of patients carrying a mutation in the LMNA gene.

In order to identify these factors that modulate the clinical severity of laminopathies, the investigators wish to collect biological material (muscle and/or skin biopsies) from patients carrying a mutation in the LMNA gene. The study of this biological material using multi OMICs technics will allow the investigators to identify and functionally validate the action of these modifying genes.

OMIICs is a set of techniques for characterising biological molecules using high-throughput approaches such as DNA sequencing, RNA sequencing and/or chromatin conformation (ATACseq...), proteins.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an LMNA mutation that has led to the diagnosis of laminopathy affecting striated muscle
* Presenting the symptoms of the disease, whether they are index cases or related to this index case (muscle weakness, tendon retractions with or without respiratory or cardiac involvement)
* Have no contraindication to muscle or skin biopsy, i.e., 1) presence of a history of allergy to latex, antiseptics, local anesthetics and adhesive dressings, 2) Current oral or parenteral anticoagulant therapy (anti-vitamin K, heparins, anti-platelet agents, anti-factor X, anti-thrombin), 3) History of inherited (haemophilias, platelet diseases) or acquired (vitamin K deficiency, liver failure) coagulation disorders.
* Patients (adult participant) or both holders of parental authority (minor participant) must sign a free and informed consent. If a minor has only 1 legal representative, the latter must attest to this on the consent form.
* Patients affiliated to the general French social security system, to the French Universal Medical Coverage (CMU) or to any French equivalent scheme.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Adult subject to legal protection measures (safeguard of justice, curatorship and guardianship).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle severity outcome | 5 years
  Will be a composite scale combining maximal motor acquisitions (sitting, walking, running) and what remains as motor skills with disease course (still running, only walking, only sitting, inability to sit)). In details:
  * The maximal motor acquisitions (M2A) : no motor acquisitions = 0, only rolling = 1, only sitting = 2, only walking = 3, running = 4.
  * The remaining motor skills (RMS) with disease course: still running = 3, only walking = 2, only sitting = 1, inability to sit = 0.
  The composite scale for a given patient will be M2A + RMS.
Cardiac muscle severity outcome | 5 years
  Will be a composite scale according to left ventricle ejection fraction (normal>55%, moderate <55% and >45%, severe<45%) and the presence or absence of conduction defects and arrhythmias.
Protective structural variant outcome | 5 years
  Structural gene variants identified on patient biological materials by Whole Genome Sequencing (WGS), associated with the mild disease severity.
Protective differential gene expression outcome | 5 years
  differential gene expression identified on patient biological materials by RNA sequencing (RNA-seq) associated with the mild disease severity.
Protective 3D chromatin conformation outcome | 5 years
  3D conformation of chromatin identified on patient biological materials by Chromatin Immuno-Precipitaiton Sequencing (CHIP Seq) associated with the mild disease severity.
Aggravating structural variant outcome | 5 years
  Structural gene variants identified on patient biological materials by Whole Genome Sequencing (WGS), associated with the worse disease severity.
Aggravating differential gene expression outcome | 5 years
  Differential gene expression identified on patient biological materials by RNA sequencing (RNA-seq) associated with the worse disease severity.
Aggravating 3D chromatin conformation outcome outcome | 5 years
  3D conformation of chromatin identified on patient biological materials by Chromatin Immuno-Precipitaiton Sequencing (CHIP Seq) associated with the worse disease severity.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Centre de référence maladies neuromusculaires, Hôpital Femme Mère Enfant, CHU Lyon, Bron, Auvergne-Rhône-Alpes
  - Service de Neuropédiatrie, Centre de Référence Maladies Neuromusculaires, CHU de Montpellier, Montpellier, Hérault
  - Service de Génétique médicale, CHU Rennes, Rennes, Ille-et-Vilaine
  - Laboratoire d'Explorations Fonctionnelles - Centre de Référence Maladies Neuromusculaires Rares, CHU Nantes, Nantes, Loire-Atlantique
  - Service de cardiologie & Service de Neurophysiologie - CHU de Rouen, Rouen, Normandy
  - Centre de référence maladies neuromusculaires, Institut de myologie, Hôpital Pitié-Salpêtrière, Paris
  - Centre de référence pour les maladies cardiaques héréditaires, Paris
  - Service de Neurologie, Réanimation Pédiatriques, Hôpital Raymond Poincaré, Hôpitaux Universitaires, Paris-Ile-de-France-Ouest, Garches, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Granger B, Gueneau L, Drouin-Garraud V, Pedergnana V, Gagnon F, Ben Yaou R, Tezenas du Montcel S, Bonne G. Modifier locus of the skeletal muscle involvement in Emery-Dreifuss muscular dystrophy. Hum Genet. 2011 Feb;129(2):149-59. doi: 10.1007/s00439-010-0909-1. Epub 2010 Nov 10. PMID 21063730
- [Background] Ben Yaou R, Yun P, Dabaj I, Norato G, Donkervoort S, Xiong H, Nascimento A, Maggi L, Sarkozy A, Monges S, Bertoli M, Komaki H, Mayer M, Mercuri E, Zanoteli E, Castiglioni C, Marini-Bettolo C, D'Amico A, Deconinck N, Desguerre I, Erazo-Torricelli R, Gurgel-Giannetti J, Ishiyama A, Kleinsteuber KS, Lagrue E, Laugel V, Mercier S, Messina S, Politano L, Ryan MM, Sabouraud P, Schara U, Siciliano G, Vercelli L, Voit T, Yoon G, Alvarez R, Muntoni F, Pierson TM, Gomez-Andres D, Reghan Foley A, Quijano-Roy S, Bonnemann CG, Bonne G. International retrospective natural history study of LMNA-related congenital muscular dystrophy. Brain Commun. 2021 Apr 11;3(3):fcab075. doi: 10.1093/braincomms/fcab075. eCollection 2021 Jul. PMID 34240052
- See also: UMD LMNA mutation database — http://www.umd.be/LMNA/